CLINICAL TRIAL: NCT06463236
Title: Clinical Validation of the Management Process for Renal Anemia in Maintenance Hemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Daqing (Other)
Responsible Party: Sponsor-Investigator, Hong Daqing, Chief physician, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Anemia of Chronic Kidney Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Standardized guidance for anemia treatment by grassroots doctors using the maintenance hemodialysis renal anemia management process
  Interventions: Other: Guiding treatment
- control group (Active Comparator): Experiential treatment by grassroots doctors
  Interventions: Other: empirical therapy

INTERVENTIONS:
Other: Guiding treatment — Standardized guidance for anemia treatment by grassroots doctors using the maintenance hemodialysis renal anemia management process
  Arms: Intervention group
Other: empirical therapy — Experiential treatment by grassroots doctors
  Arms: control group

SUMMARY:
This test aims to verify that the management process of renal anemia in maintenance hemodialysis patients can improve the hemoglobin compliance rate better than that of anemia management by primary doctors, and promote the system at the grassroots level to guide primary doctors in anemia management and improve the management standard of renal anemia in maintenance hemodialysis patients through prospective randomized controlled trials. To improve the anemia compliance rate of maintenance hemodialysis patients, and to improve the basic doctors' grasp of the anemia management guidelines, consensus and standard operating procedures.

ELIGIBILITY:
Inclusion Criteria:

① Age over 18 years old; ② Receive regular hemodialysis at least twice a week for at least 3 months, and have no plans to stop hemodialysis within 6 months since the start of the trial; ③ The patient voluntarily participated in this study.

Exclusion Criteria:

* Patients who have planned to undergo kidney transplantation or terminate hemodialysis during the study period; ② Previous history of bone marrow hematopoietic system diseases, such as combined myelodysplastic syndrome, multiple myeloma, and other diseases; ③ Any known hereditary blood disease, such as thalassemia, sickle cell anemia, pure red blood cell aplasia, etc.; ④ Active or chronic gastrointestinal bleeding; ⑤ There was a severe infection within one week prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1296 (Estimated)
Dates: Start 2024-06-14 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the one-year compliance rate of renal anemia | one year
  Changes in renal anemia compliance rates between the experimental group and the control group within one year

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided